CLINICAL TRIAL: NCT00004194
Title: A Phase I-II Study for the Treatment of Steroid Resistant GVHD With Fludarabine
Brief Title: Fludarabine in Treating Patients With Steroid-Resistant Chronic Graft- Versus-Host Disease
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Supportive Care
Other Study IDs: CDR0000067435; UCLA-9701029; NCI-G99-1650
Record Dates: First submitted 2000-01-21; First posted 2004-09-16 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2000-04

CONDITIONS: Graft Versus Host Disease
Keywords: graft versus host disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — fludarabine phosphate

INTERVENTIONS:
Drug: fludarabine phosphate

SUMMARY:
RATIONALE: Fludarabine may be an effective treatment for graft-versus-host disease caused by bone marrow transplantation.

PURPOSE: Phase I/II trial to study the effectiveness of fludarabine in treating patients who have chronic graft-versus-host disease that has not responded to steroid therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose, toxicity, and efficacy of fludarabine in patients with steroid resistant chronic graft versus host disease.

OUTLINE: This is a dose escalation study. Phase I: Patients receive fludarabine IV over less than 30 minutes for 1-3 days. Treatment repeats every 4 weeks for up to 4 courses in the absence of relapse of underlying disease, malignancy, graft rejection, or unacceptable toxicity. Patients with progressive graft versus host disease after completion of 3 courses are taken off study. Patients with complete response are taken off study. Patients with partial response may continue treatment at the immediate prior dose level. Cohorts 3-6 patients receive escalating doses of fludarabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 3 of 6 patients experience dose limiting toxicity. Phase II: Patients receive fludarabine at the MTD from phase I of the study.

PROJECTED ACCRUAL: A total of 15-27 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or clinically proven chronic graft versus host disease (GVHD) that has failed to respond to at least 1 month of treatment with the following: Steroids (greater than 0.5 mg/kg/day) AND Cyclosporine or a cytotoxic agent (azathioprine or mercaptopurine) OR Other experimental treatment (such as chloroquine) All allogeneic bone marrow or peripheral blood stem cell transplantation patients eligible regardless of underlying disease for which transplantation was performed if: At least 45 days since prior transplantation No relapse of underlying disease No loss of donor hematopoiesis Patients with a rapid deterioration of GVHD that is considered life threatening if not controlled are eligible after receiving high dose steroids (greater than 1 mg/kg/day) for at least 10 days

PATIENT CHARACTERISTICS: Age: Not specified Performance status: Not specified Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,300/mm3 Platelet count at least 75,000/mm3 Hepatic: Not specified Renal: Creatinine no greater than 2 mg/dL Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics Chemotherapy: No other concurrent cytotoxic drugs Endocrine therapy: Concurrent steroids allowed but must be tapered to less than 0.5 mg/kg/day of prednisone or equivalent prior to starting study drug (if symptomatic flare develops during taper, patients may continue on the lowest dose thought to produce stabilization) Radiotherapy: Not specified Surgery: Not specified Other: Concurrent cyclosporine and other nonmyelosuppressive drugs allowed No concurrent myelosuppressive agents (azathioprine, mercaptopurine)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Christos E. Emmanouilides, MD, Study Chair — Jonsson Comprehensive Cancer Center